CLINICAL TRIAL: NCT07047053
Title: Evaluation of the Anti-VZV Vaccine Response of Patients With Immune-mediated Systemic Inflammatory Diseases Vaccinated in the Care Setting
Acronym: ZONAMID
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP250443; 2025-A00547-42 (Other: IDRCB)
Record Dates: First submitted 2025-06-19; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Vaccination Varicella-zoster Virus; Immune-mediated Systemic Inflammatory Diseases
Keywords: varicella-zoster virus; vaccination
MeSH Terms: conditions — Chickenpox

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with immune-mediated systemic inflammatory diseases (IMID): All patients treated for IMID in the internal medicine department of Hôpital Bichat, vaccinated against VZV as part of their care, in accordance with HAS recommendations.

SUMMARY:
Patients with immune-mediated systemic inflammatory diseases (IMID) are at increased risk of shingles due to treatment-induced immunosuppression. In line with international recommendations, the French National Authority for Health (HAS) updated the varicella-zoster virus (VZV) vaccination strategy in March 2024. The HAS now recommends that immunocompromised people aged 18 and over be vaccinated with the recombinant VZV vaccine. However, due to the immunosuppressive treatment received, the vaccine response in MIMI patients is often suboptimal, and the protection induced by the herpes zoster vaccine in this context is unknown.

The aim of our study is to determine the rate of anti-VZV seroconversion after vaccination with recombinant anti-VZV vaccine, in patients followed up for MIMI.

DETAILED DESCRIPTION:
Vaccination with the recombinant anti-VZV vaccine (Shingrix) is carried out as part of treatment in all immunocompromised patients over 18 years of age, in accordance with HAS recommendations (the vaccination schedule requires 2 doses 2 months apart).

The vaccine response will be measured during hospitalisation and/or follow-up consultations, using the same sample as that used to monitor MIMI in the same laboratory (Immunology Laboratory, CHU Bichat).

Clinical and biological data will be collected to study factors associated with vaccine response, vaccine tolerance and MIMI activity.

Information relating to diagnosis, examinations and follow-up will be collated in the patient's medical file.

Patients are systematically seen every 6 months for follow-up consultations as part of their MIMI.

No additional visits are planned for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age being managed for MIMI, including
* Systemic lupus
* Gougerot-Sjögren's syndrome
* Systemic scleroderma
* Mixed connectivitis
* Inflammatory myositis
* Systemic sarcoidosis
* Systemic vasculitis (necrotizing vasculitis and giant cell arteritis)
* Behçet's disease
* Adult Still's disease
* IgG4-associated disease
* Autoimmune cytopenias (autoimmune hemolytic anemia, immunological thrombocytopenic purpura, Evans syndrome)
* Susac syndrome
* Followed in the internal medicine department of Hôpital Bichat, Paris
* Justifying VZV vaccination due to immunosuppression or age over 65.
* Vaccinated as part of care between June 2025 and June 2026
* Regardless of history of shingles
* With a serum sample available for analysis
* Having received at least the first dose of the vaccine regimen (in hospital or in the community)

Exclusion Criteria:

* Evolving cancer, with or without treatment (chemotherapy, immunotherapy, etc.)
* History of VZV vaccination (live or recombinant)
* Patient who has had an allergic reaction to a vaccine
* Pregnancy
* Patient under legal protection, guardianship or trusteeship
* Not affiliated to a social security scheme (general or CMU)
* Patient unable to understand research information
* Absence of non-opposition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated for IMID in the internal medicine department of Hôpital Bichat, vaccinated against VZV as part of their care, in accordance with HAS recommendations.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Levels of antibodies specific to VZV gE glycoprotein and levels of specific T lymphocytes after stimulation with peptides contained in the vaccine (in SFC/106 PBMC) | at 3 and/or 6 month
level of antibodies specific to the VZV gE glycoprotein after stimulation with peptides contained in the vaccine (in SFC/106 PBMC) | at 3 and/or 6 month

SECONDARY OUTCOMES:
Frequency of specific T cells | before vaccination, at 3 and/or 6 month
Tolerance of the VZV vaccine | at 3 and/or 6 month
  occurrence of non-serious adverse events
Safety of the VZV vaccine | at 3 and/or 6 month
  occurrence of serious adverse events
measuring change in IMID (Immune mediated inflammatory disease) activity. The data collected will be aggregated into a composite score. | at 3 and/or 6 month
  The measures used depend on the scale specific to each IMID. The parameters collected will be the scales (SLEDAI for SLE, ESSDAI for Sjögren's syndrome, mRSS for systemic sclerosis, BSAS for Behcet's disease and BVAS for vasculitis), the physiological parameters collected by the referring doctor and, where appropriate, certain biological activity parameters (C-reactive protein, anti-DNA, ANCA, etc.). The data collected will be aggregated into a composite score.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Bichat, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided